CLINICAL TRIAL: NCT06715670
Title: A Phase I, Randomized, Open-label, Single-dose, Four-period, Four-treatment, Cross-over Study to Assess the Pharmacokinetics of Zibotentan in Healthy Non-Asian and Japanese Participants
Brief Title: A Study to Investigate the Blood Concentrations of 4 Different Oral Doses of Zibotentan in Healthy Non-Asian and Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D4326C00010
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Liver Cirrhosis
Keywords: Chronic kidney disease; Treatment sequence; Pharmacokinetics; Washout periods
MeSH Terms: conditions — Liver Cirrhosis; Renal Insufficiency, Chronic | interventions — ZD4054

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment sequence ABCD: Zibotentan (Experimental): Participants will receive single dose of Zibotentan in 4 occassions with first Treatment A, followed by Treatment B, Treatment C and then Treatment D with each dose separated by 3 washout periods.
  Interventions: Drug: Zibotentan
- Treatment sequence BDAC: Zibotentan (Experimental): Participants will receive single dose of Zibotentan in 4 occassions with first Treatment B, followed by Treatment D, Treatment A and then Treatment C with each dose separated by 3 washout periods
  Interventions: Drug: Zibotentan
- Treatment sequence CADB: Zibotentan (Experimental): Participants will receive single dose of Zibotentan in 4 occassions with first Treatment C, followed by Treatment A, Treatment D and then Treatment B with each dose separated by 3 washout periods.
  Interventions: Drug: Zibotentan
- Treatment sequence DCBA: Zibotentan (Experimental): Participants will receive single dose of Zibotentan in 4 occassions with first Treatment D, followed by Treatment C, Treatment B and then Treatment A with each dose separated by 3 washout periods.
  Interventions: Drug: Zibotentan

INTERVENTIONS:
Drug: Zibotentan — Participant will receive 4 different single doses of zibotentan on Day 1 of each treatment period orally.

SUMMARY:
This study aim to assess the Pharmacokinetics of Zibotentan in Healthy Non-Asian and Japanese Participants.

DETAILED DESCRIPTION:
This study will be Phase I, randomized, open-label, single-dose, 4-period, 4-treatment, cross-over study, performed at a single study center.

The study will comprise: Screening Period of maximum 28 days; Four Treatment Periods, separated by 3 washout periods; Final Follow-up Visit within 5 to 7 days after the last study intervention administration. The washout periods will last at least 3 days, resulting in a total dosing-free time of at least 6 full days between each of the 4 treatments. Participant will receive the first dose is on Day 1, then the next dose will be on Day 8 at the earliest.

Each participant will receive 4 different single doses (Dose 1, 2, 3 and 4) of zibotentan, at all 4 studied dose levels in one of the following treatment sequences: ABCD, BDAC, CADB, DCBA.

Each participant will be involved in the study for approximately 9 weeks, depending upon the duration of the washout periods.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male and female (non-childbearing potential) with suitable veins for cannulation or repeated venipuncture.
* All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit.
* Females of non-childbearing potential must be confirmed at the Screening Visit.
* Sexually active fertile male participants with partners of childbearing potential must adhere to the contraception methods.
* Body mass index (BMI) between 18 and 32 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive at Screening.
* Japanese participant must have Japanese parents and grandparents, were born in Japan, and not have lived outside Japan for over 10 years.
* Participant is considered non-Asian if their parents and all grandparents are ethnically non-Asian.

Exclusion Criteria:

* History of any clinically important disease or disorder which may either put the participant at risk because of participation in the study or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* Any clinically important abnormalities in clinical chemistry, hematology, or urinalysis, laboratory values and vital signs at the Screening Visit.
* Any positive result on Screening for serum HBsAg (Hepatitis B surface antigen), HBcAb (Hepatitis B core antibody) or HIV (Human immunodeficiency virus).
* Clinically significant abnormal findings in vital signs after 10 minutes of supine rest.
* Clinically important abnormalities in rhythm, conduction, or morphology of the resting electrocardiography (ECG) and prolonged QTcF > 450 ms, family history of long QT syndrome, or early cardiac death.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
* Positive screen for drugs of abuse or alcohol at Screening or first admission.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity.
* Excessive intake of caffeine-containing drinks or food.
* Use of any prescribed or nonprescribed medication, including antacids, analgesics, herbal remedies, mega dose vitamins, and minerals within 2 weeks before the first administration of the study intervention.
* Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months before the Screening Visit.
* Receipt of another new chemical entity within 30 days or 5 half-lives (whichever is longest) of the first administration of the study intervention.
* Previous receipt of zibotentan within 28 days before Day 1 dosing in the Clinical Unit.
* Treatment with strong or moderate Cytochrome P450 3A4 (CYP3A4) inhibitors or inducers within 28 days or 5 half-lives (whichever is longest) or weak CYP3A4 inhibitors or inducers within 3 days or 3 half-lives (whichever is longest) before dosing.
* Involvement in the planning and/or conduct of the study.
* Ongoing or recent minor medical complaints that may interfere with the interpretation of study data or compliance with study procedures.
* Being vegan or having medical dietary restrictions.
* Inability to communicate reliably with the Principal Investigator or designee.
* Being a vulnerable participant, such as those kept in detention, under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Area under concentration-time curve from time 0 to infinity (AUCinf) | Day 1 through Day 3 of each Treatment Period (each Treatment Period is 7 days)
  To characterize the single-dose plasma PK of orally administered zibotentan in healthy non-Asian and Japanese participants.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | Day 1 through Day 3 of each Treatment Period (each Treatment Period is 7 days)
  To characterize the single-dose plasma PK of orally administered zibotentan in healthy non-Asian and Japanese participants.
Maximum observed drug concentration (Cmax) | Day 1 through Day 3 of each Treatment Period (each Treatment Period is 7 days)
  To characterize the single-dose plasma PK of orally administered zibotentan in healthy non-Asian and Japanese participants

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) receiving single dose | From Screening (28 days) to follow-up Visit 5 to 7 days post-final dose (approximately 9 weeks)
  To assess the safety and tolerability of receiving single dose of orally administered zibotentan.
Concentration at 24 hours post dose (C24) | Day 1 through Day 3 of each Treatment Period (each Treatment Period is 7 days)
  To further characterize zibotentan PK in plasma.
Partial area under the concentration time curve from time 0 to 24 hours post-dose (AUC(0-24)) | Day 1 through Day 3 of each Treatment Period (each Treatment Period is 7 days)
  To further characterize zibotentan PK in plasma.
Time to reach maximum observed concentration (tmax) | Day 1 through Day 3 of each Treatment Period (each Treatment Period is 7 days)
  To further characterize zibotentan PK in plasma.
Terminal elimination half-life (t1/2 λz) | Day 1 through Day 3 of each Treatment Period (each Treatment Period is 7 days)
  To further characterize zibotentan PK in plasma.
Mean residence time (MRTinf) | Day 1 through Day 3 of each Treatment Period (each Treatment Period is 7 days)
  To further characterize zibotentan PK in plasma.
Terminal rate constant (λz) | Day 1 through Day 3 of each Treatment Period (each Treatment Period is 7 days)
  To further characterize zibotentan PK in plasma.
Apparent total body clearance (CL/F) | Day 1 through Day 3 of each Treatment Period (each Treatment Period is 7 days)
  To further characterize zibotentan PK in plasma.
Apparent volume of distribution based on the terminal phase (Vz/F) | Day 1 through Day 3 of each Treatment Period (each Treatment Period is 7 days)
  To further characterize zibotentan PK in plasma.
Individual and cumulative amount of unchanged drug excreted into urine (Ae) (by time point and cumulative) | Day 1 through Day 3 of each Treatment Period (each Treatment Period is 7 days)
  To further characterize zibotentan PK in urine.
Individual and cumulative percentage of dose excreted unchanged in urine from time t1 to time t2 (fe) (by time point and cumulative) | Day 1 through Day 3 of each Treatment Period (each Treatment Period is 7 days)
  To further characterize zibotentan PK in urine.
Renal clearance (CLR) | Day 1 through Day 3 of each Treatment Period (each Treatment Period is 7 days)
  To further characterize zibotentan PK in urine.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/